CLINICAL TRIAL: NCT04728061
Title: A Phase 1a/1b, Randomized, Double-blind, Placebo-Controlled, Single and Multiple Ascending Dose Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of GEn1E-1124 After Single and Multiple IV Infusion Dosing in Healthy Volunteers
Brief Title: Study to Assess the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of GEn1E-1124
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GEn1E Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GEn1E-1124-001
Record Dates: First submitted 2021-01-22; First posted 2021-01-28 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Ascending Dose (Experimental)
  Interventions: Drug: Gen1E-1124; Drug: Placebo
- Multiple Ascending Dose (Experimental)
  Interventions: Drug: Gen1E-1124; Drug: Placebo

INTERVENTIONS:
Drug: Gen1E-1124 — Intravenously-infused Gen1E-1124 in vehicle.
Drug: Placebo — Intravenously-infused vehicle.

SUMMARY:
In this early phase clinical research study, the investigational drug will be administered to 64 healthy volunteers in a double-blind, placebo-controlled manner, at a one research center. The objectives of the study are to assess what the body does to the investigational drug, what the investigational drug does to the body and also to observe the safety and tolerability of the investigational drug healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects;
2. Between 18 and 55 years of age;
3. Provide a signed EC-approved consent form;
4. Generally healthy, in the opinion of the Investigator;
5. Body Mass Index (BMI) 18 to 30 kg/m^2;
6. Creatinine clearance with in specific parameter;
7. Using method of contraception;
8. Willing and able to comply with protocol requirements for the duration of the study.

Exclusion Criteria:

1. Subjects taking prohibited medication;
2. Subjects with a history or presence of clinically significant medical or psychiatric disease;
3. Subjects who have regularly used nicotine-containing products ;
4. Subjects who have used caffeine-containing products;
5. Subjects who are unable to comply with eating a standardized meal during the study;
6. Subjects with a hospital admission or major surgery within 30 days prior to Screening;
7. Subjects with a plasma donation within 7 days prior to Screening;
8. Subjects who have not abstained from alcoholic beverages/alcohol-containing products at least 72 hours prior to first dose, or plan to consume them at any time through completion of the Follow-up Visit;
9. Subjects who cannot refrain from strenuous exercise from 72 hours prior to dose administration through completion of the Follow-up Visit;
10. Subjects who are pregnant or breastfeeding
11. Subjects who have participated (taken investigative drug and/or device) in another clinical trial within 90 days prior to Screening;
12. Subjects who are employees of the study unit or their family members, students who are working in the study unit, or family members of the Investigator or Sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-06-18 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events from the start of randomization through the final follow-up visit | Up to 14 days post-dose

SECONDARY OUTCOMES:
Plasma levels of GEn1E-1124 and potential metabolites | Through 24 hours post-dose
Urine levels of GEn1E-1124 and potential metabolites | Through 24 hours post-dose
Cytokines measured in whole blood | Up to 24 hours post-dose
Selected biomarkers measured in whole blood | Up to 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Lal, PhD, MS, Study Director — GEn1E Lifesciences
Locations (1):
- GEn1E-1124 Clinical Research Site, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — https://www.gen1elifesci.com/